CLINICAL TRIAL: NCT03979469
Title: Criteria Based Discharge in Ambulatory Surgery in Children Undergoing Opioid Versus Opioid Free Anesthesia
Brief Title: Opioid Versus Non-opioid Anesthesia for Ambulatory Surgery in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athens General Children's Hospital "Pan. & Aglaia Kyriakou" (Other)
Responsible Party: Principal Investigator, Adelais Tsiotou, Consultant of Anesthesiology Department, Athens General Children's Hospital "Pan. & Aglaia Kyriakou"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Opioid free anesthesia 7.2018
Record Dates: First submitted 2019-05-09; First posted 2019-06-07 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Effect of Anesthesia in Postoperative Pain; Effect of Anesthesia in Extubation Time; Effect of Anesthesia in Discharge Time From Postanesthesia Care Unit; Effect of Anesthesia in Postoperative Adverse Events; Effect of Anesthesia in Discharge Time From the Hospital
MeSH Terms: interventions — Ketamine; Dexmedetomidine; Fentanyl; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- opiod free general anesthesia (Experimental): In group A opioid free anesthesia is administered. Anesthesia and analgesia were achieved with ketamine(1mg/kg, bolus), dexmedetomidine(1mcg/kg, over 10 minutes), local anesthetic(ropivacaine 2mg/kg 0.75% wound infiltration), paracetamol(15mg/kg), non steroid analgesics(diclofenac 1mg/kg). Anesthesia induction with ketamine(1mg/kg), propofol 1% 2-3mg/kg, rocuronium 1mg/kg. Anesthesia maintenance with propofol 1% 10mg/kg/hour. Reversal of rocuronium with sugammadex 2mg/kg.
  Interventions: Drug: Ketamine, dexmedetomidine
- opioid based general anesthesia (Active Comparator): In group B opioid based anesthesia is administered.Anesthesia and analgesia were achieved with remifentanil(0.3mcg/kg/minute), local anesthetic(ropivacaine 2mg/kg 0.75% wound infiltration), paracetamol(15mg/kg), non steroid analgesics(diclofenac 1mg/kg).Anesthesia induction with propofol 1% 2-3mg/kg,fentanyl(2mcg/kg), rocuronium 1mg/kg. Anesthesia maintenance with propofol 1% 10mg/kg/hour. Reversal of rocuronium with sugammadex 2mg/kg.
  Interventions: Drug: fentanyl, remifentanil

INTERVENTIONS:
Drug: Ketamine, dexmedetomidine — Patients will receive non-opioid analgesics, such as dexmedetomidine, ketamine perioperatively
  Arms: opiod free general anesthesia
Drug: fentanyl, remifentanil — Patients will receive opioid analgesics, such as fentanyl and remifentanil perioperatively
  Arms: opioid based general anesthesia

SUMMARY:
The investigators intend to study the safety and effectiveness of opioid free anesthesia compared to opioid anesthesia in ambulatory surgery in children, regarding postoperative pain, hemodynamic stability, agitation and discharge times. Quality of postanesthetic care was estimated in a 24h follow up.

ELIGIBILITY:
Inclusion Criteria:

* children,
* American Society Anesthesia I, II,
* ambulatory surgery

Exclusion Criteria:

* Allergy to anesthetic and analgesic drugs,
* history of neuromuscular,
* renal, neurological, hepatic disease,
* craniofacial anomalies,
* Obstructive Sleep Apnea,
* obesity,
* cardiopulmonary diseases

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Discharge times from the hospital | 4 hours
  Comparison of the discharge times from the hospital between opioid free and opioid based anesthesia using Discharge criteria based on physiological scoring system, evaluating respiration, circulation, level of consciousness, postoperative pain, postoperative nausea and vomiting and surgical site. A score 12 or more allows patient to leave safely from the hospital.
Severity of postoperative pain | 24 hours
  Comparison of the severity of postoperative pain between opioid free and opioid based anesthesia using Visual Analogue Scale for children aged 7 years and more. We instruct the patient to point to the position on the line between the faces to indicate how much pain they are currently feeling. The far left end indicates "no pain"(0) and the far right end indicates "worst pain ever."(10)
Severity of postoperative pain | 24 hours
  Comparison of the severity of postoperative pain between opioid free and opioid based anesthesia using the Face, Legs, Activity, Cry, Consolability scale or FLACC scale for children between the ages of 3 years and 7 years. The scale has five criteria, which are each assigned a score of 0, 1 or 2.The scale is scored in a range of 0-10 with 0 representing no pain.

SECONDARY OUTCOMES:
Extubation time | 30 minutes
  Comparison of extubation time, time interval between discontinuation of anesthetics and extubation between the two groups
Discharge time from PACU | 60 minutes
  Comparison of discharge time from postanesthesia unit, time interval between arrival from operating room until leaving postanesthesia unit, between the two groups using Aldrete scale, score of 9 or greater allows patient to leave postanesthesia unit
Cost effect | 24 hours
  Comparison of hospitalization fees among the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital P. and A. Kyriakou Anesthesiology Department, Athens, Greece

IPD SHARING:
Plan to Share IPD: No